CLINICAL TRIAL: NCT00860782
Title: Parent Intervention to Improve Academic Success in Children With Sickle Cell Disease
Brief Title: Parent Educational Program for Children With Sickle Cell Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Daniel F. Armstrong, Professor of Pediatrics, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20080278; U54HL090569 (NIH); U54HL090569-01 (NIH)
Record Dates: First submitted 2009-03-10; First posted 2009-03-12 (Estimated); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Hemoglobin SC Disease; Anemia, Sickle Cell
Keywords: Sickle Cell Disease; Educational Outcomes; Neurodevelopmental Functioning
MeSH Terms: conditions — Hemoglobin SC Disease; Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Annual Parent Intervention (API) Group (Experimental): Participants in this group will receive the parent educational support intervention once a year for 2 years.
  Interventions: Behavioral: Parent Educational Support
- Quarterly Parent Intervention (QPI) Group (Experimental): Participants in this group will receive the parent educational support intervention quarterly (4 times a year) for 2 years.
  Interventions: Behavioral: Parent Educational Support

INTERVENTIONS:
Behavioral: Parent Educational Support — Parents will attend 45-minute educational sessions that will focus on providing them with information regarding SCD and how they can best help their child perform better in school.

SUMMARY:
Children with sickle cell disease (SCD) are at risk for central nervous system (CNS) complications, which may affect academic achievement. This study will evaluate an educational support program for parents that aims to improve academic achievement in children with SCD.

DETAILED DESCRIPTION:
SCD is an inherited blood disorder that is caused by an abnormal type of hemoglobin-the protein in red blood cells that carries oxygen to tissues. Symptoms include anemia, infections, organ damage, and intense episodes of pain, which are called "sickle cell crises." Children with SCD are also at risk for a variety of CNS complications, including various types of stroke and increased blood flow to the brain. These conditions affect neuropsychological performance and academic achievement. In children with SCD, there may also be a relationship between CNS complications, behavioral problems, family environment stressors, and pain symptoms. For example, children with SCD-related CNS complications have a higher risk of developing behavioral problems than children without SCD. In turn, behavioral problems are associated with high levels of family conflict and can be a significant stressor for families coping with SCD. This kind of stress can then lead to increased difficulty in dealing with SCD symptoms, particularly pain, for the child. This study will evaluate an educational support program for parents of children with SCD, conducted either once a year or four times a year, in terms of the program's effect on children's academic achievement. In addition, study researchers will also evaluate the program's effect on behavioral difficulties, pain frequency, and the family environment.

This study will enroll children with HbSS (sickle cell anemia) or HbSb-thal (hemoglobin S beta thalassemia) SCD. Parents or caregivers of participants will be randomly assigned to attend the educational support program meetings either once a year or four times a year for 2 years. The educational meetings with the parent/caregiver will be 45 minutes long and will cover the following four main areas:

1. Provide education regarding the learning issues often seen with children with SCD
2. Provide information regarding special education services in the school system and how the parent can obtain academic support for his/her child
3. Provide information on how to assist the child to better manage homework
4. Evaluate the child's current level of pain and how pain may affect school attendance

There will be three evaluation timepoints. At baseline and Year 3, children will undergo a neurodevelopmental evaluation, including academic achievement tests. The parent and child will complete questionnaires on emotional and behavioral functioning, stress levels, and family functioning. At Year 2, the children will complete academic achievement tests, and the questionnaires for the parent and child will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Children with either HbSS (sickle cell anemia) or HbSβ-thal (hemoglobin S beta thalassemia) who are between 6 and 12 years of age
* Child's parent or primary caregiver agrees to participate in the study

Exclusion Criteria:

* Child is monolingual in a language other than English and cannot complete standardized testing in English
* Parent or caregiver of the child is not fluent in English or Spanish
* Child has some other developmental disability not related to SCD. This would include Down's syndrome, autism, pervasive developmental disability, cerebral palsy, seizure disorder, consequences of severe prematurity, or a documented closed head injury that resulted in loss of consciousness.
* Child has been diagnosed with a significant mental health disorder that is not responsive to behavioral or medical management. This includes severe depression, schizophrenia, or bipolar disorder. Children whose mental health problem is effectively treated are eligible for participation.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Academic achievement as measured by the Woodcock Johnson Tests of Achievement, Third Edition | Measured at baseline and Years 2 and 3
  Performance on standardized measure of academic achievement, M=100, SD=15

SECONDARY OUTCOMES:
Child's emotional and behavioral functioning, parental stress, and family functioning | Measured at baseline and Years 2 and 3
  Standardized parent report quesionnaires of child adjustment, parent stress, and family function

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Armstrong, PhD, Study Director — University of Miami
Locations (1):
- Mailman Center for Child Development, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Following final data analysis and dissemination, the SAP and ICF will be shared with investigators requesting these materials.